CLINICAL TRIAL: NCT06162507
Title: A Multicenter, Single-arm, Open-label Study to Evaluate the Safety, Pharmacokinetics, and Pharmacokinetics of CM310 in Children Subjects With Moderate-to-severe Atopic Dermatitis
Brief Title: Study of CM310 in Children Subjects With Moderate-to-severe Atopic Dermatis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Keymed Biosciences Co.Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CM310-101010
Record Dates: First submitted 2023-11-29; First posted 2023-12-08 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2023-11

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CM310 group A (Experimental): CM310 injection, subcutaneous injection, once every 3 weeks.
  Interventions: Biological: CM310
- CM310 group B (Experimental): CM310 injection, subcutaneous injection, once every 2 weeks.
  Interventions: Biological: CM310

INTERVENTIONS:
Biological: CM310 — CM310 injection

SUMMARY:
This is a multi-center, single arm, open-label study to evaluate safety in children patients with moderate-to severe atopic dermatis.

ELIGIBILITY:
Inclusion Criteria:

* With atopic dermatis.
* Voluntarily sign the informed consent form.

Exclusion Criteria:

* Any major surgery planned during the research period.
* With intestinal parasitic infection within the first 6 months of screening.
* With any previous malignant tumors prior to screening.
* With any circumstance that is not suitable to participate in this study.

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2023-12-22 (Actual); Primary Completion 2024-07-04 (Actual); Study Completion 2024-07-04 (Actual)

PRIMARY OUTCOMES:
Adverse events | up to week 16
  Incidence of adverse events.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Children's Hospital Capital Medical University, Beijing, China